CLINICAL TRIAL: NCT00221559
Title: Serum Zn Status of Patients With Cystic Fibrosis at Diagnosis and One Year Later, Compared to a Healthy Control Group
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Scientific research fund Bruges (Unknown)
Other Study IDs: UZGhent 001
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Blood sampling for determination of serum Zn

SUMMARY:
Serum Zn status of patients with cystic fibrosis at diagnosis and one year later, compared to a healthy control group

DETAILED DESCRIPTION:
Serum Zn status of patients with cystic fibrosis at diagnosis and one year later, compared to a healthy control group

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Van Biervliet, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Result] Van Biervliet S, Van Biervliet JP, Robberecht E. Serum zinc in patients with cystic fibrosis at diagnosis and after one year of therapy. Biol Trace Elem Res. 2006 Sep;112(3):205-11. doi: 10.1385/BTER:112:3:205. PMID 17057259
- See also: Website University Hospital Ghent — http://www.uzgent.be